CLINICAL TRIAL: NCT03920488
Title: Evaluating the Feasibility of Next-Generation Sequencing - Based Germline and Somatic Genetic Testing in Triple-negative Breast Cancer. The PERSONA-breast Trial
Brief Title: Next-Generation Sequencing-based Germline and Somatic Genetic Testing in Triple-negative Breast Cancer
Acronym: PERSONA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0761/
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Triple Negative Breast Cancer
Keywords: genetic testing; breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients with triple negative breast cancer, implementation of genetic testing in decision making might impact both risk management for the patient and her family, but also, importantly, therapeutic management.

Identifying genetically predisposed subjects dictates risk-reducing strategies that may imply bilateral salpingo-oophorectomy and mastectomy or long term medical approaches. In the advanced setting, genetic testing can influence decision for medical therapy (e.g. use of platinum derivatives, poly-ADP ribose polymerase inhibitors (PARP inhibitors) in breast cancer patients with breast cancer susceptibility gene (BRCA) mutation.

The selection of patients for testing has long relied on the presence of a strong family history of breast and ovarian cancer. It is now clear that this criterion will result in substantial numbers of those with a BRCA mutation being missed.

Systematic large-scale genetic testing, simultaneously on germline and somatic tissues, is likely to improve decisional algorithms in patients with ovarian cancer. Feasibility of such approach in the clinical setting, in terms of a turnaround time compatible with clinical needs and sensitivity comparable if not superior to single-gene testing needs to be demonstrated before such diagnostic platforms can be routinely implemented in the diagnostic workflow. This is the scope of the present study.

DETAILED DESCRIPTION:
Systematic large-scale genetic testing, simultaneously on germline and somatic tissues, is likely to improve decisional algorithms in patients with triple negative breast cancers.

Feasibility of such approach in the clinical setting, in terms of a turnaround time compatible with clinical needs and sensitivity comparable if not superior to single-gene testing needs to be demonstrated before such diagnostc platforms can be routinely implemented in the diagnostic workflow.

Two platforms will be used during the course of the study. The Illumina TruSight Cancer Risk panel is a commercially validated targeted enrichment panel which targets 94 genes and 284 SNPs (Single Nucleotide Polymorphism) associated with a predisposition towards cancer.

The GermSom panel was developed at European Institute of Oncology (IEO) in collaboration with institutions within the Alleanza Contro il Cancro consortium and manufactured by Agilent Technologies. It includes 349 genes with an established function in the biology and/or pharmacological actionability of multiple solid tumors, including breast cancer. It includes all the genomic regions analysed in the Illumina Trusight panel, plus 32 additional regions associated with risk of multiple tumors.

Patients will receive detailed genetic characterization of their germline and their tumor. This will provide the best possible characterization of their risk of developing of a secondary malignancy and can be exploited to identify families at risk for hereditary cancer risk. Patients will also benefit from an increased likelihood of being treated with appropriate drugs and of receiving appropriate surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 60 years
2. has signed informed consent
3. histologically confirmed triple negative breast cancer (ER (Estrogen Receptors) < 1%, PgR (Progesterone Receptors) < 1%, HER2/neu negative (IHC 0, 1+ or 2+ FISH negative).
4. Stage I-III
5. Able to undergo surgery (primary or post-neoadjuvant)
6. Availability of surgical/bioptic material within 6 months from enrolment

Exclusion Criteria:

* unable or unwilling to receive genetic counselling

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with triple-negative breast cancer, stage I-III, cadidates for surgery
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mutations in breast cancer risk-associated genes | 3 months
  Evaluate the prevalence of clinically relevant mutations in breast cancer risk-associated genes
Genetic test turnaround time | 6 months
  Evaluate feasibility of genetic testing for clinical decision making
Percentage of informative specimens | 3 months
  Percentage of patients with positive germline testing for target genes

SECONDARY OUTCOMES:
Incidence of all other mutations | 3 months
  Incidence of all other mutations
disease-free survival | 10 years
  collection of disease associated events during follow-up
overall survival | 10 years
  collection of death events during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Viviana E Galimberti, MD, Principal Investigator — IEO
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy

IPD SHARING:
Plan to Share IPD: No